CLINICAL TRIAL: NCT05269615
Title: Exercise-induced Erythropoiesis: the Mechanistic of Angiotensin II
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19200831
Record Dates: First submitted 2022-02-04; First posted 2022-03-08 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-12

CONDITIONS: Exercise Physiology
MeSH Terms: interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be randomly allocated in a 1:1 ratio to valsartan or placebo. Valsartan and placebo tablets will be indistinguishable in taste, smell, appearance and dosage. The protocol will be developed in a double-blind manner in that both participants and investigators will be blinded toward the intervention condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Valsartan tablets (Active Comparator)
  Interventions: Drug: Valsartan 80 mg
- Placebo tablets (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valsartan 80 mg — The well-established angiotensin II receptor blocker (ARB) valsartan will be used in the present study to selectively block AT1 receptors. Valsartan is a generic medication widely used in hypertensive patients since 1996 as well as safely applied in physiological studies comprising healthy individuals.1-3 A minimal valsartan dose of 80 mg known to acutely reduce circulating EPO levels in healthy individuals will be provided 4 hours before starting Study 1 to optimize AT1 blockade according to valsartan's half-life.1-3 The same dose of valsartan (80 mg) will be provided 4 hours before each ET session in Study 2. The participants will be randomly allocated in a 1:1 ratio to valsartan or placebo. Valsartan and placebo tablets will be indistinguishable in taste, smell, appearance and dosage. The protocol will be developed in a double-blind manner in that both participants and investigators will be blinded toward the intervention condition.
  Arms: Valsartan tablets
Drug: Placebo — The participants will be randomly allocated in a 1:1 ratio to valsartan or placebo. Valsartan and placebo tablets will be indistinguishable in taste and smell. The protocol will be developed in a double-blind manner in that both participants and investigators will be blinded toward the intervention condition.
  Arms: Placebo tablets

SUMMARY:
The major aims are to determine the effect of acute (single dose) blockade of ANGII receptor 1 (AT1) on the EPO response to a single session of endurance exercise, as well as determine the effect of chronic (8-week) blockade of AT1 on ET-induced adaptations in total circulating red blood volume and hemoglobin.

DETAILED DESCRIPTION:
Physical activity, particularly when comprised of endurance training (ET) leading to cardiovascular adaptations, is considered the most effective intervention to augment life expectancy. Major health benefits induced by ET are closely associated (independently of traditional risk factors) with improvements in maximal oxygen consumption (VO2max), a hallmark of aerobic exercise capacity. The higher the VO2max the greater the likelihood to be free of cardiovascular disease, the main cause of mortality worldwide. Understanding the mechanisms explaining the improvement in VO2max with ET can provide sound basis for highly effective lifestyle and pharmacological interventions aimed to enhance cardiovascular health in the general population. So far, the essential role of ET-induced increased formation of red blood cells, i.e., erythropoiesis, has been firmly established for any improvement in VO2max. Yet, the underlying mechanism remains elusive. Clinical studies and recent investigations by the PI point towards the endocrine effects of key hormones that regulate blood volume (BV). Notably, the impact of ET-induced changes in angiotensin II (ANGII), a multifaceted hormone that modulates erythropoiesis through its effects on kidney erythropoietin (EPO) production, has to be experimentally elucidated in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status, absence of current medical symptoms or medication limiting incremental exercise testing
* No history of cardiac, pulmonary or kidney disease.

Exclusion Criteria:

- Individuals fulfilling the above criteria but currently involved in regular exercise training (> 5 hr/week)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
stroke volume in ml/m2 | 10 weeks
  Stroke volume (SV) will be determined as left ventricular end-diastolic volume (LVEDV) minus left ventricular end-systolic volume (LVESV)
maximal oxygen consumption in ml/kg/min | 10 weeks
  Maximal oxygen consumption (VO2max), a hallmark of aerobic capacity, will be determined with continuous measurements of oxgyen uptake using an online gas collection system (Quark CPET, Cosmed, Italy)
Blood volume (BV)-regulating hormone: Plasma ANGII in ng/dL | 10 weeks
  Plasma ANGII concentrations will be quantified by means of established competitive enzyme immunoassays

CONTACTS AND LOCATIONS:
Locations (1):
- School of Public Health, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided